CLINICAL TRIAL: NCT02766712
Title: The Physiological Effects of Pacing on Catheter Ablation Procedures to Treat Atrial Fibrillation
Acronym: PEP AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 16-00813
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CA 1st Half of lesion (Experimental): During each of the 15 pre-specified lesions, pacing will be initiated at a 500ms cycle length from a catheter in the coronary sinus or right ventricle prior to the start of the lesion. Pacing will be stopped at the halfway point (e.g. after 10 seconds for a 20-second lesion and after 15 seconds for a 30-second lesion). In the event that Wenckebach behavior is noted, pacing will be adjusted to a 550ms cycle length. In the event that Wenckebach behavior persists, the cycle length will be adjusted to 600ms. In the event that Weckebach behavior continues, the pacing catheter will be moved to the right ventricle, which and pacing will be performed at a 500ms cycle length. If Wenckebach behavior still persists, the patient will be withdrawn from the study.
  Interventions: Procedure: Pace During 1st Half of Lesion
- CA 2nd Half of Lesion (Experimental): During each of the 15 pre-specified lesions, pacing will be stopped at the halfway point (e.g. after 10 seconds for a 20-second lesion and after 15 seconds for a 30-second lesion). In the event that Wenckebach behavior is noted, pacing will be adjusted to a 550ms cycle length. In the event that Wenckebach behavior persists, the cycle length will be adjusted to 600ms. In the event that Wenckebach behavior persists, the pacing catheter will be moved to the right ventricle and pacing will be performed at a 500ms cycle length. If Wenckebach behavior still persists, the patient will be withdrawn from the study.
  Interventions: Procedure: Pace During 2nd Half of Lesion

INTERVENTIONS:
Procedure: Pace During 1st Half of Lesion
  Arms: CA 1st Half of lesion
Procedure: Pace During 2nd Half of Lesion
  Arms: CA 2nd Half of Lesion

SUMMARY:
This is a two arm randomized, paired prospective study comparing the percentage of time spent above Contact Force (CF), Force Time Integral (FTI) and other lesion parameters in the setting of pacing versus non-pacing. This study is designed to compare the percentage of time spent above CF 10 grams between paced and non-paced lesions at 15 pre-determined lesion locations.

DETAILED DESCRIPTION:
Patients will be randomized and proceed to one of two study arms:

1. Pacing during first half of lesions: During each of the 15 pre-specified lesions, pacing will be initiated at a 500ms cycle length from a catheter in the coronary sinus or right ventricle prior to the start of the lesion. Pacing will be stopped at the halfway point (e.g. after 10 seconds for a 20-second lesion and after 15 seconds for a 30-second lesion). In the event that Wenckebach behavior is noted, pacing will be adjusted to a 550ms cycle length. In the event that Wenckebach behavior persists, the cycle length will be adjusted to 600ms. In the event that Weckebach behavior continues, the pacing catheter will be moved to the right ventricle, which and pacing will be performed at a 500ms cycle length. If Wenckebach behavior still persists, the patient will be withdrawn from the study.
2. Pacing during second half of lesions: During each of the 15 pre-specified lesions, pacing will be stopped at the halfway point (e.g. after 10 seconds for a 20-second lesion and after 15 seconds for a 30-second lesion). In the event that Wenckebach behavior is noted, pacing will be adjusted to a 550ms cycle length. In the event that Wenckebach behavior persists, the cycle length will be adjusted to 600ms. In the event that Wenckebach behavior persists, the pacing catheter will be moved to the right ventricle and pacing will be performed at a 500ms cycle length. If Wenckebach behavior still persists, the patient will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AF scheduled for AF ablation with planned pulmonary vein isolation
* Presenting in normal sinus rhythm (NSR) prior to lesion delivery

Exclusion Criteria:

* Previous radiofrequency ablation
* Previous thoracotomy-type AF ablation (MAZE or similar technique)
* In AF prior to lesion delivery
* Evidence of left atrial scarring on voltage map
* Resting heart rate > 90 bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Left superior pulmonary vein | 20 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Left middle pulmonary vein | 20 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Left inferior pulmonary vein | 20 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Right superior pulmonary | 20 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Right middle pulmonary vein | 20 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Right inferior pulmonary vein | 20 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Left superior pulmonary vein | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Left pulmonary vein carina | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Left inferior pulmonary vein | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Right superior pulmonary | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Right pulmonary vein carina | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Right inferior pulmonary vein | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Anterior CTI | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Middle CTI | 30 Seconds
Percentage of time spent above CF 10 grams between paced and non-paced lesions at Posterior CTI | 30 Seconds

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Aizer, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aizer A, Cheng AV, Wu PB, Qiu JK, Barbhaiya CR, Fowler SJ, Bernstein SA, Park DS, Holmes DS, Chinitz LA. Pacing Mediated Heart Rate Acceleration Improves Catheter Stability and Enhances Markers for Lesion Delivery in Human Atria During Atrial Fibrillation Ablation. JACC Clin Electrophysiol. 2018 Apr;4(4):483-490. doi: 10.1016/j.jacep.2017.12.017. Epub 2018 Mar 1. PMID 30067488